CLINICAL TRIAL: NCT00072995
Title: Preventing Overweight Using Novel Dietary Strategies (Pounds Lost)
Brief Title: Preventing Obesity Using Novel Dietary Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank M. Sacks, Professor of Medicine, Brigham and Women's Hospital
Purpose: Prevention
Other Study IDs: 1238; U01HL073286 (NIH)
Record Dates: First submitted 2003-11-13; First posted 2003-11-17 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Fatty Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Four Diets Differing in Macronutrient Composition
Behavioral: Diets Low in Saturated Fat

SUMMARY:
The purpose of this study is to test the effectiveness for weight loss and weight maintenance of four diets differing in macronutrient composition: moderate in fat (40 percent energy) with two different protein levels (15 percent and 25 percent), and low in fat (20 percent energy), also with 15 percent and 25 percent protein levels. The study is only accepting participants in the Boston, Massachusetts or Baton Rouge, Louisiana area. For further enrollment information in Boston or Baton Rouge, see Eligibility Criteria or Design Narrative.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity is a growing problem whose importance is reflected in the resources that are expended each year by a large section of the population on weight reduction drugs and therapies. Although numerous weight loss diets are available, there is little agreement in the scientific literature or the lay press as to the amount of fat, protein, and carbohydrates that would comprise the most efficacious diet for weight loss and long term weight loss retention. Reliable information about the effectiveness of low calorie diets with differing macronutrient composition is clearly needed and of paramount importance to inform the choice of a weight reduction diet.

DESIGN NARRATIVE:

The study tests the effectiveness for weight loss and weight maintenance of four diets differing in macronutrient composition: moderate in fat (40% energy) with two different protein levels (15% and 25%), and low in fat (20% energy), also with 15% and 25% protein levels. The moderate-fat diet will be patterned after a Mediterranean diet. All four dietary approaches will be low in saturated fat, and will involve reduction in total energy intake. Each diet is deemed practical and suitable for public health recommendations, and each would be expected to have a favorable effect on cardiovascular disease risk factors. All participants will receive a state-of-the-art behavioral therapy program standardized across the two centers in Boston and Baton Rouge. An estimated 800 men and women, age 30-70 years, body mass index (BMI) 25-40 kg/m2, will be randomized among the 4 dietary treatments. The primary outcome variable will be change in total body weight from baseline to 2 years. Secondary outcomes related to obesity are body fat, BMI, waist circumference, visceral fat, and hepatic and skeletal muscle fat. Other outcomes are psychological factors (diet satisfaction, satiety, food craving, dietary restraint, disinhibition and hunger, and quality of life); major cardiovascular risk factors (blood pressure, low density lipoprotein [LDL] cholesterol, high density lipoprotein [HDL] cholesterol, and triglycerides); prevalence of the metabolic syndrome; blood glucose, insulin, and hemoglobin A1C; emerging cardiovascular risk factors (apolipoprotein B, VLDL and LDL particles with apolipoprotein C-III, lipoprotein[a]); microalbuminuria; and bone mineral content. The primary results will be straightforwardly applicable to public health and clinical guidelines for obesity and will increase our understanding of the biology of obesity and weight loss.

The study is only accepting participants in the Boston, Massachusetts or Baton Rouge, Louisiana area. For Boston participants, contact: 617-998-1047 or www.poundslost.org. For Baton Rouge participants, contact: schoensj@pbrc.edu or 225-763-2623.

ELIGIBILITY:
Inclusion Criteria:

* Only accepting participants in the Boston, Massachusetts or Baton Rouge, Louisiana area
* Between the ages of 30 - 70
* Willing to modify eating pattern according to instructions
* Overweight or obese and in good health with a BMI of 25-40
* Committed to a long-term weight loss and maintenance program
* Willing to attend multiple weight loss group sessions
* Willing to increase activity level

Exclusion Criteria:

* Pregnant, planning to become pregnant, or are breastfeeding
* Unwilling to participate in the schedule of group sessions and individual visits
* Unstable or recent onset of heart disease or any other serious illness
* Cannot change diet due to medical or other reasons
* Planning to leave the area prior to the anticipated end of participation
* Current participation in another clinical trial with an intervention that affects weight change
* Have diabetes that is treated with insulin or hypoglycemic oral medicines
* Diagnosis of psychiatric or emotional problems within 6 months of study
* Currently have an eating disorder
* Have hypothyroidism
* Have an unstable weight

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811
Dates: Start 2003-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight (measured at Year 2)

SECONDARY OUTCOMES:
Body fat
BMI
Waist circumference
Visceral fat
Hepatic and skeletal muscle
Psychological factors from diet
Major cardiovascular risk factors
Prevalence of the metabolic syndrome (measured at Year 2)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pennington Biomedical Reseach Center, Louisiana State University, Baton Rouge, Louisiana
  - Harvard University School of Public Health, Boston, Massachusetts

REFERENCES:
- [Derived] Heianza Y, Xue Q, Rood J, Clish CB, Bray GA, Sacks FM, Qi L. Changes in bile acid subtypes and improvements in lipid metabolism and atherosclerotic cardiovascular disease risk: the Preventing Overweight Using Novel Dietary Strategies (POUNDS Lost) trial. Am J Clin Nutr. 2024 May;119(5):1293-1300. doi: 10.1016/j.ajcnut.2024.02.019. Epub 2024 Feb 28. PMID 38428740
- [Derived] Xue Q, Heianza Y, Li X, Wang X, Ma H, Rood J, Dorans KS, Mills KT, Liu X, Bray GA, Sacks FM, Qi L. Circulating MicroRNA-19 and cardiovascular risk reduction in response to weight-loss diets. Clin Nutr. 2024 Mar;43(3):892-899. doi: 10.1016/j.clnu.2024.02.015. Epub 2024 Feb 15. PMID 38382419
- [Derived] Heianza Y, Xue Q, Rood J, Bray GA, Sacks FM, Qi L. Circulating thrifty microRNA is related to insulin sensitivity, adiposity, and energy metabolism in adults with overweight and obesity: the POUNDS Lost trial. Am J Clin Nutr. 2023 Jan;117(1):121-129. doi: 10.1016/j.ajcnut.2022.10.001. Epub 2022 Dec 15. PMID 36789931
- [Derived] Li A, Li X, Zhou T, Ma H, Heianza Y, Williamson DA, Smith SR, Bray GA, Sacks FM, Qi L. Sleep Disturbance and Changes in Energy Intake and Body Composition During Weight Loss in the POUNDS Lost Trial. Diabetes. 2022 May 1;71(5):934-944. doi: 10.2337/db21-0699. PMID 35202470
- [Derived] Heianza Y, Zhou T, He H, DiDonato JA, Bray GA, Sacks FM, Qi L. Changes in gut-microbiota-related metabolites and long-term improvements in lipoprotein subspecies in overweight and obese adults: the POUNDS lost trial. Int J Obes (Lond). 2021 Dec;45(12):2600-2607. doi: 10.1038/s41366-021-00939-7. Epub 2021 Aug 23. PMID 34426648
- [Derived] Han L, Zhang T, You D, Chen W, Bray G, Sacks F, Qi L. Temporal and mediation relations of weight loss, and changes in insulin resistance and blood pressure in response to 2-year weight-loss diet interventions: the POUNDS Lost trial. Eur J Nutr. 2022 Feb;61(1):269-275. doi: 10.1007/s00394-021-02643-8. Epub 2021 Jul 28. PMID 34319427
- [Derived] Li X, Sun D, Zhou T, Ma H, Heianza Y, Liang Z, Bray GA, Sacks FM, Qi L. Changes of Branched-Chain Amino Acids and Ectopic Fat in Response to Weight-loss Diets: the POUNDS Lost Trial. J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3747-56. doi: 10.1210/clinem/dgaa377. PMID 32561903
- [Derived] Heianza Y, Zhou T, Yuhang C, Huang T, Willett WC, Hu FB, Bray GA, Sacks FM, Qi L. Starch Digestion-Related Amylase Genetic Variants, Diet, and Changes in Adiposity: Analyses in Prospective Cohort Studies and a Randomized Dietary Intervention. Diabetes. 2020 Sep;69(9):1917-1926. doi: 10.2337/db19-1257. Epub 2020 Jun 3. PMID 32493715
- [Derived] Chen Y, Zhou T, Sun D, Li X, Ma H, Liang Z, Heianza Y, Pei X, Bray GA, Sacks FM, Qi L. Distinct genetic subtypes of adiposity and glycemic changes in response to weight-loss diet intervention: the POUNDS Lost trial. Eur J Nutr. 2021 Feb;60(1):249-258. doi: 10.1007/s00394-020-02244-x. Epub 2020 Apr 9. PMID 32274554
- [Derived] Liu X, Hanseman DJ, Champagne CM, Bray GA, Qi L, Williamson DA, Anton SD, Sacks FM, Tong J. Predicting Weight Loss Using Psychological and Behavioral Factors: The POUNDS LOST Trial. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1274-83. doi: 10.1210/clinem/dgz236. PMID 31802116
- [Derived] Sun D, Zhou T, Li X, Heianza Y, Liang Z, Bray GA, Sacks FM, Qi L. Genetic Susceptibility, Dietary Protein Intake, and Changes of Blood Pressure: The POUNDS Lost Trial. Hypertension. 2019 Dec;74(6):1460-1467. doi: 10.1161/HYPERTENSIONAHA.119.13510. Epub 2019 Oct 28. PMID 31656094
- [Derived] Zhou T, Heianza Y, Chen Y, Li X, Sun D, DiDonato JA, Pei X, LeBoff MS, Bray GA, Sacks FM, Qi L. Circulating Gut Microbiota Metabolite Trimethylamine N-Oxide (TMAO) and Changes in Bone Density in Response to Weight Loss Diets: The POUNDS Lost Trial. Diabetes Care. 2019 Aug;42(8):1365-1371. doi: 10.2337/dc19-0134. Epub 2019 May 21. PMID 31332027
- [Derived] Miketinas DC, Bray GA, Beyl RA, Ryan DH, Sacks FM, Champagne CM. Fiber Intake Predicts Weight Loss and Dietary Adherence in Adults Consuming Calorie-Restricted Diets: The POUNDS Lost (Preventing Overweight Using Novel Dietary Strategies) Study. J Nutr. 2019 Oct 1;149(10):1742-1748. doi: 10.1093/jn/nxz117. PMID 31174214
- [Derived] Heianza Y, Sun D, Li X, DiDonato JA, Bray GA, Sacks FM, Qi L. Gut microbiota metabolites, amino acid metabolites and improvements in insulin sensitivity and glucose metabolism: the POUNDS Lost trial. Gut. 2019 Feb;68(2):263-270. doi: 10.1136/gutjnl-2018-316155. Epub 2018 Jun 2. PMID 29860242
- [Derived] Liu G, Dhana K, Furtado JD, Rood J, Zong G, Liang L, Qi L, Bray GA, DeJonge L, Coull B, Grandjean P, Sun Q. Perfluoroalkyl substances and changes in body weight and resting metabolic rate in response to weight-loss diets: A prospective study. PLoS Med. 2018 Feb 13;15(2):e1002502. doi: 10.1371/journal.pmed.1002502. eCollection 2018 Feb. PMID 29438414
- [Derived] Heianza Y, Sun D, Smith SR, Bray GA, Sacks FM, Qi L. Changes in Gut Microbiota-Related Metabolites and Long-term Successful Weight Loss in Response to Weight-Loss Diets: The POUNDS Lost Trial. Diabetes Care. 2018 Mar;41(3):413-419. doi: 10.2337/dc17-2108. Epub 2018 Jan 5. PMID 29305401
- [Derived] Han L, Ma W, Sun D, Heianza Y, Wang T, Zheng Y, Huang T, Duan D, Bray JGA, Champagne CM, Sacks FM, Qi L. Genetic variation of habitual coffee consumption and glycemic changes in response to weight-loss diet intervention: the Preventing Overweight Using Novel Dietary Strategies (POUNDS LOST) trial. Am J Clin Nutr. 2017 Nov;106(5):1321-1326. doi: 10.3945/ajcn.117.156232. Epub 2017 Sep 20. PMID 28931532
- [Derived] Heianza Y, Sun D, Wang T, Huang T, Bray GA, Sacks FM, Qi L. Starch Digestion-Related Amylase Genetic Variant Affects 2-Year Changes in Adiposity in Response to Weight-Loss Diets: The POUNDS Lost Trial. Diabetes. 2017 Sep;66(9):2416-2423. doi: 10.2337/db16-1482. Epub 2017 Jun 28. PMID 28659346
- [Derived] Apolzan JW, Myers CA, Champagne CM, Beyl RA, Raynor HA, Anton SA, Williamson DA, Sacks FM, Bray GA, Martin CK. Frequency of Consuming Foods Predicts Changes in Cravings for Those Foods During Weight Loss: The POUNDS Lost Study. Obesity (Silver Spring). 2017 Aug;25(8):1343-1348. doi: 10.1002/oby.21895. Epub 2017 Jun 15. PMID 28618170
- [Derived] Huang T, Zheng Y, Hruby A, Williamson DA, Bray GA, Shen Y, Sacks FM, Qi L. Dietary Protein Modifies the Effect of the MC4R Genotype on 2-Year Changes in Appetite and Food Craving: The POUNDS Lost Trial. J Nutr. 2017 Mar;147(3):439-444. doi: 10.3945/jn.116.242958. Epub 2017 Feb 1. PMID 28148682
- [Derived] Ma W, Huang T, Heianza Y, Wang T, Sun D, Tong J, Williamson DA, Bray GA, Sacks FM, Qi L. Genetic Variations of Circulating Adiponectin Levels Modulate Changes in Appetite in Response to Weight-Loss Diets. J Clin Endocrinol Metab. 2017 Jan 1;102(1):316-325. doi: 10.1210/jc.2016-2909. PMID 27841942
- [Derived] Heianza Y, Ma W, Huang T, Wang T, Zheng Y, Smith SR, Bray GA, Sacks FM, Qi L. Macronutrient Intake-Associated FGF21 Genotype Modifies Effects of Weight-Loss Diets on 2-Year Changes of Central Adiposity and Body Composition: The POUNDS Lost Trial. Diabetes Care. 2016 Nov;39(11):1909-1914. doi: 10.2337/dc16-1111. Epub 2016 Aug 31. PMID 27581055
- [Derived] Vadiveloo M, Sacks FM, Champagne CM, Bray GA, Mattei J. Greater Healthful Dietary Variety Is Associated with Greater 2-Year Changes in Weight and Adiposity in the Preventing Overweight Using Novel Dietary Strategies (POUNDS Lost) Trial. J Nutr. 2016 Aug;146(8):1552-9. doi: 10.3945/jn.115.224683. Epub 2016 Jun 29. PMID 27358422
- [Derived] Huang T, Ley SH, Zheng Y, Wang T, Bray GA, Sacks FM, Qi L. Genetic susceptibility to diabetes and long-term improvement of insulin resistance and beta cell function during weight loss: the Preventing Overweight Using Novel Dietary Strategies (POUNDS LOST) trial. Am J Clin Nutr. 2016 Jul;104(1):198-204. doi: 10.3945/ajcn.115.121186. Epub 2016 Jun 8. PMID 27281308
- [Derived] Wang T, Huang T, Zheng Y, Rood J, Bray GA, Sacks FM, Qi L. Genetic variation of fasting glucose and changes in glycemia in response to 2-year weight-loss diet intervention: the POUNDS LOST trial. Int J Obes (Lond). 2016 Jul;40(7):1164-9. doi: 10.1038/ijo.2016.41. Epub 2016 Mar 22. PMID 27113490
- [Derived] Zheng Y, Ceglarek U, Huang T, Li L, Rood J, Ryan DH, Bray GA, Sacks FM, Schwarzfuchs D, Thiery J, Shai I, Qi L. Weight-loss diets and 2-y changes in circulating amino acids in 2 randomized intervention trials. Am J Clin Nutr. 2016 Feb;103(2):505-11. doi: 10.3945/ajcn.115.117689. Epub 2016 Jan 20. PMID 26791187
- [Derived] Qi Q, Zheng Y, Huang T, Rood J, Bray GA, Sacks FM, Qi L. Vitamin D metabolism-related genetic variants, dietary protein intake and improvement of insulin resistance in a 2 year weight-loss trial: POUNDS Lost. Diabetologia. 2015 Dec;58(12):2791-9. doi: 10.1007/s00125-015-3750-1. Epub 2015 Sep 29. PMID 26416604
- [Derived] Lin X, Qi Q, Zheng Y, Huang T, Lathrop M, Zelenika D, Bray GA, Sacks FM, Liang L, Qi L. Neuropeptide Y genotype, central obesity, and abdominal fat distribution: the POUNDS LOST trial. Am J Clin Nutr. 2015 Aug;102(2):514-9. doi: 10.3945/ajcn.115.107276. Epub 2015 Jul 8. PMID 26156739
- [Derived] Xu M, Ng SS, Bray GA, Ryan DH, Sacks FM, Ning G, Qi L. Dietary Fat Intake Modifies the Effect of a Common Variant in the LIPC Gene on Changes in Serum Lipid Concentrations during a Long-Term Weight-Loss Intervention Trial. J Nutr. 2015 Jun;145(6):1289-94. doi: 10.3945/jn.115.212514. Epub 2015 Apr 29. PMID 25926410
- [Derived] Tirosh A, de Souza RJ, Sacks F, Bray GA, Smith SR, LeBoff MS. Sex Differences in the Effects of Weight Loss Diets on Bone Mineral Density and Body Composition: POUNDS LOST Trial. J Clin Endocrinol Metab. 2015 Jun;100(6):2463-71. doi: 10.1210/jc.2015-1050. Epub 2015 Mar 31. PMID 25825948
- [Derived] Zheng Y, Huang T, Zhang X, Rood J, Bray GA, Sacks FM, Qi L. Dietary Fat Modifies the Effects of FTO Genotype on Changes in Insulin Sensitivity. J Nutr. 2015 May;145(5):977-82. doi: 10.3945/jn.115.210005. Epub 2015 Mar 11. PMID 25761503
- [Derived] Thomas DM, Ivanescu AE, Martin CK, Heymsfield SB, Marshall K, Bodrato VE, Williamson DA, Anton SD, Sacks FM, Ryan D, Bray GA. Predicting successful long-term weight loss from short-term weight-loss outcomes: new insights from a dynamic energy balance model (the POUNDS Lost study). Am J Clin Nutr. 2015 Mar;101(3):449-54. doi: 10.3945/ajcn.114.091520. Epub 2014 Dec 24. PMID 25733628
- [Derived] Huang T, Huang J, Qi Q, Li Y, Bray GA, Rood J, Sacks FM, Qi L. PCSK7 genotype modifies effect of a weight-loss diet on 2-year changes of insulin resistance: the POUNDS LOST trial. Diabetes Care. 2015 Mar;38(3):439-44. doi: 10.2337/dc14-0473. Epub 2014 Dec 12. PMID 25504030
- [Derived] Huang T, Qi Q, Li Y, Hu FB, Bray GA, Sacks FM, Williamson DA, Qi L. FTO genotype, dietary protein, and change in appetite: the Preventing Overweight Using Novel Dietary Strategies trial. Am J Clin Nutr. 2014 May;99(5):1126-30. doi: 10.3945/ajcn.113.082164. Epub 2014 Mar 12. PMID 24622803
- [Derived] Mirzaei K, Xu M, Qi Q, de Jonge L, Bray GA, Sacks F, Qi L. Variants in glucose- and circadian rhythm-related genes affect the response of energy expenditure to weight-loss diets: the POUNDS LOST Trial. Am J Clin Nutr. 2014 Feb;99(2):392-9. doi: 10.3945/ajcn.113.072066. Epub 2013 Dec 11. PMID 24335056
- [Derived] Nicklas JM, Sacks FM, Smith SR, LeBoff MS, Rood JC, Bray GA, Ridker PM. Effect of dietary composition of weight loss diets on high-sensitivity c-reactive protein: the Randomized POUNDS LOST trial. Obesity (Silver Spring). 2013 Apr;21(4):681-9. doi: 10.1002/oby.20072. PMID 23712970
- [Derived] Xu M, Qi Q, Liang J, Bray GA, Hu FB, Sacks FM, Qi L. Genetic determinant for amino acid metabolites and changes in body weight and insulin resistance in response to weight-loss diets: the Preventing Overweight Using Novel Dietary Strategies (POUNDS LOST) trial. Circulation. 2013 Mar 26;127(12):1283-9. doi: 10.1161/CIRCULATIONAHA.112.000586. Epub 2013 Feb 27. PMID 23446828
- [Derived] Mattei J, Qi Q, Hu FB, Sacks FM, Qi L. TCF7L2 genetic variants modulate the effect of dietary fat intake on changes in body composition during a weight-loss intervention. Am J Clin Nutr. 2012 Nov;96(5):1129-36. doi: 10.3945/ajcn.112.038125. Epub 2012 Oct 3. PMID 23034957
- [Derived] Zhang X, Qi Q, Bray GA, Hu FB, Sacks FM, Qi L. APOA5 genotype modulates 2-y changes in lipid profile in response to weight-loss diet intervention: the Pounds Lost Trial. Am J Clin Nutr. 2012 Oct;96(4):917-22. doi: 10.3945/ajcn.112.040907. Epub 2012 Aug 22. PMID 22914552
- [Derived] de Souza RJ, Bray GA, Carey VJ, Hall KD, LeBoff MS, Loria CM, Laranjo NM, Sacks FM, Smith SR. Effects of 4 weight-loss diets differing in fat, protein, and carbohydrate on fat mass, lean mass, visceral adipose tissue, and hepatic fat: results from the POUNDS LOST trial. Am J Clin Nutr. 2012 Mar;95(3):614-25. doi: 10.3945/ajcn.111.026328. Epub 2012 Jan 18. PMID 22258266
- [Derived] Qi Q, Bray GA, Hu FB, Sacks FM, Qi L. Weight-loss diets modify glucose-dependent insulinotropic polypeptide receptor rs2287019 genotype effects on changes in body weight, fasting glucose, and insulin resistance: the Preventing Overweight Using Novel Dietary Strategies trial. Am J Clin Nutr. 2012 Feb;95(2):506-13. doi: 10.3945/ajcn.111.025270. Epub 2012 Jan 11. PMID 22237064
- [Derived] Qi Q, Bray GA, Smith SR, Hu FB, Sacks FM, Qi L. Insulin receptor substrate 1 gene variation modifies insulin resistance response to weight-loss diets in a 2-year randomized trial: the Preventing Overweight Using Novel Dietary Strategies (POUNDS LOST) trial. Circulation. 2011 Aug 2;124(5):563-71. doi: 10.1161/CIRCULATIONAHA.111.025767. Epub 2011 Jul 11. PMID 21747052
- [Derived] Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, McManus K, Champagne CM, Bishop LM, Laranjo N, Leboff MS, Rood JC, de Jonge L, Greenway FL, Loria CM, Obarzanek E, Williamson DA. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009 Feb 26;360(9):859-73. doi: 10.1056/NEJMoa0804748. PMID 19246357